CLINICAL TRIAL: NCT03710707
Title: A Phase 1b, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL201 in Subjects With Parkinson's Disease
Brief Title: Study to Evaluate DNL201 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-B-0002
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: LRRK2; Parkinson's Disease; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — 2-methyl-2-(3-methyl-4-((4-(methylamino)-5-(trifluoromethyl)pyrimidin-2-yl)amino)-1H-pyrazol-1-yl)propanenitrile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DNL201 low dose (Experimental)
  Interventions: Drug: DNL201
- DNL201 high dose (Experimental)
  Interventions: Drug: DNL201
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL201 — Oral repeating dose
  Arms: DNL201 high dose; DNL201 low dose
Drug: Placebo — Oral repeating dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple oral doses of DNL201 in subjects with Parkinson's disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) between 18 and 35.0 kg/m2, inclusive
* Clinical diagnosis of Parkinson's disease meeting UK Brain Bank criteria and H&Y Stage I, II, or III.
* sPD subgroup without a LRRK2 mutation; PD LRRK2 subgroup with LRRK2 mutation
* Screening dopamine transporter (DAT) SPECT scan with a DAT deficit consistent with Parkinson's disease
* Able to hold Parkinson's disease medications 8 hours (overnight) prior to specific study assessments

Key Exclusion Criteria:

* Any history of clinically significant asthma, chronic obstructive pulmonary disease, or emphysema within 5 years of screening, or other clinically significant pulmonary disease within 6 months of screening
* Abnormal Vitals including Respiratory Rate, Body Temperature, and Blood Pressure
* Pulmonary Function Tests (PFTs) (FVC <60% predicted, FEV1 <50% predicted, FEV1:FVC ratio <0.6, DLCO <70% predicted)
* Clinically significant neurologic disorder other than Parkinson's disease, including history of stroke, cognitive impairment, seizure within 5 years of screening, or head trauma with loss of consciousness within 6 months of screening
* Montreal Cognitive Assessment (MoCA) score of <24 at screening

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Randomization to Day 42
Number of Subjects with laboratory test abnormalities | Randomization to Day 42
Number of Subjects with vital sign abnormalities | Randomization to Day 42
Number of Subjects with electrocardiogram (ECG) abnormalities | Randomization to Day 42
Number of Subjects with clinically significant neurological examination abnormalities | Randomization to Day 42

SECONDARY OUTCOMES:
Pharmacokinetic measure of maximum observed plasma concentration (Cmax) of DNL201 | Randomization to Day 28
Pharmacokinetic measure of time to reach maximum observed plasma concentration (Tmax) of DNL201 | Randomization to Day 28
Pharmacokinetic measure of trough plasma observed concentration (Ctrough) of DNL201 | Randomization to Day 28
Pharmacokinetic measure of area under the plasma drug concentration-time curve (AUC) of DNL201 | Randomization to Day 28
Pharmacokinetic measure of CSF concentrations of DNL201 | Randomization to Day 28
Pharmacodynamic measure of pS935 in whole blood and/or PBMCs | Randomization to Day 28
Pharmacodynamic measure of pRab10 in PBMCs | Randomization to Day 28

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Clinical Site(s), Long Beach, California
  - Clinical Site(s), Aurora, Colorado
  - Clinical Site(s), Miami, Florida
  - Clinical Site(s), Orlando, Florida
  - Clinical Site(s), Farmington Hills, Michigan
  - Clinical Site(s), Philadelphia, Pennsylvania
  - Clinical Site(s), Spokane, Washington

REFERENCES:
- [Derived] Maloney MT, Wang X, Ghosh R, Andrews SV, Maciuca R, Masoud ST, Agam M, Caprioli RM, Astarita G, Bondar VV, Chen J, Chiu CL, Davis SS, Ho AC, Nguyen HN, Propson NE, Reyzer ML, Davis OB, Deen MC, Zhu S, Di Paolo G, Vocadlo DJ, Estrada AA, de Vicente J, Lewcock JW, Arguello A, Suh JH, Huntwork-Rodriguez S, Henry AG. LRRK2 kinase activity regulates Parkinson's disease-relevant lipids at the lysosome. Mol Neurodegener. 2025 Aug 6;20(1):89. doi: 10.1186/s13024-025-00880-7. PMID 40770658
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102